CLINICAL TRIAL: NCT04548076
Title: Investigation of Analgesic Efficacy of Thoracolumbar Interfascial Plane Block in Vertebral Surgery
Brief Title: Thoracolumbar Interfascial Plane Block in Vertebral Surgery
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Tokat Gaziosmanpasa University, Tokat Gaziosmanpasa University
Other Study IDs: 20-KAEK-076
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Block
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Block group — Control group
  Other Names: Patients received thoracolumbar interfascial plane block before operation

SUMMARY:
To determine the postoperative analgesic efficiency of thoracolumbar interfascial plane block , patients are divided into two groups. Study group received ultrasound-guided thoracolumbar interfascial plane block , where control had none. Visual analog scale and opioid consumption are recorded.

DETAILED DESCRIPTION:
Thoracolumbar interfascial plane block has successfully been demonstrated to provide an efficient analgesia in patients. The present study is aimed to investigate the intraoperative hemodynamic responses, anesthetic and analgesic consumption, and postoperative recovery quality of thoracolumbar interfascial plane block in patients with vertebral surgery. After approval, patients enrolled in the study are divided into two groups by computer-based randomization technique as control and study group. After standard monitorization, anesthesia induction and tracheal intubation, erector spinae plane block is performed to study group and no intervention to control group.

In the intraoperative period, 10 mg / kg paracetamol and 0.05 mg / kg morphine will be used for postoperative analgesia. After surgery, all patients will be given 10 mg/kg paracetamol every 8 hours and will be fitted with a patient-controlled analgesia (PCA) device (Tramadol HCL). PCA device bolus dose will be set to 20 mg, lock time will be set to 10 minutes and the number of buttons per hour will be set as 3.for postoperative analgesia.After surgery, VAS scores of the patients will be evaluated (in the recovery room, 1,3,6,12 and 24 hours, Patients with VAS>4 will be given 0.03mg / kg morphine as salvage analgesia.After 30 minutes, the patients' VAS will be re-evaluated,If VAS>4 the same dose will be repeated. A patient satisfaction questionnaire (Qr40)will be filled by patients at the postoperative 24th hour.

ELIGIBILITY:
Inclusion Criteria:

Over 18 years of age, Planned to vertebral surgery, An American Society of Anesthesiologists score of 1,2 or 3

Exclusion Criteria:

Severe cardiovascular disease, Psychiatric diseases, Rejected to participation, Those who have chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vertebral surgery patients who will be operated under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2021-11-07 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | one time in postoperative period for one year
  Visual analog scale

SECONDARY OUTCOMES:
Opioid consumption | During postoperative period for one yea
  Opioid consumption

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tapar, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tapar H, Demir O, Genc A, Balta MG, Kolukcu V, Karaman T, Dogru S, Karaman S, Suren M. Investigation of the analgesic efficacy of ultrasound-guided thoracolumbar interfacial plane block in vertebral surgery: A prospective randomized clinical study. Saudi Med J. 2022 Oct;43(10):1136-1141. doi: 10.15537/smj.2022.43.10.20220467. PMID 36261200